CLINICAL TRIAL: NCT06487078
Title: LOREA: ANALYSIS OF THE EFFECTIVENESS AND SAFETY OF LORLATINIB IN UNTREATED ALK-POSITIVE NSCLC PATIENTS IN A FRENCH REAL-WORLD CONTEXT
Brief Title: Analysis of the Effectiveness and Safety of Lorlatinib in Untreated ALK-Positive NSCLC Patients in a French Real-World Context
Acronym: LOREA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B7461051; LOREA (Other: Alias Study Number)
Record Dates: First submitted 2024-06-05; First posted 2024-07-05 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: ALK+ Non-Small-Cell Lung Carcinoma
MeSH Terms: interventions — lorlatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lorlatinib (Experimental): Lorlatinib single agent, 100 mg (4 x 25 mg) oral tables, QD, continuously
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib — ALK-positive NSCL treatment
  Other Names: PF-06463922

SUMMARY:
Analysis of the Effectiveness and Safety of Lorlatinib in Untreated ALK-Positive NSCLC Patients in a French Real-World context

ELIGIBILITY:
Inclusion Criteria: Participants are eligible to be included in the study only if all the following criteria apply:

* Patients (male or female) 18 years of age or older at age inclusion
* Patients with histologically or cytologically confirmed diagnosis of locally advanced or metastatic (TNM 8th classification) ALK-positive NSCLC (IHC 3+/FISH positive/transcriptomic method)
* Complete radiological evaluation has to be performed before the start of lorlatinib by contrast enhanced CT-scan of thorax and upper abdomen and brain MRI, as per routine care
* Patients with ECOG performance status grade 0, 1, or 2

Exclusion Criteria: Participants are excluded from the study if any of the following criteria Apply

* Evidence of active malignancy within the last 2 years prior to inclusion (other than NSCLC, non-melanoma skin cancer, cervical in situ cancer, papillary thyroid cancer, lobular carcinoma in situ/ductal carcinoma in situ (LCIS/DCIS) of the breast, or localized prostate cancer).
* Patients who have previously received adjuvant ALK TKI therapy (unless metastatic relapse occurs more than one year after completion of adjuvant therapy).
* Patients who have previously received systemic NSCLC therapy in metastatic condition.
* Patients using any of the following food or drugs within 12 days prior to the first dose of lorlatinib:

  * known strong CYP3A inhibitors
  * known strong CYP3A inducers
  * known P gp substrates with a narrow therapeutic index
* Patients with any medical or psychiatric condition, or that may, in the investigator's judgment, increase the risk of study participation or make the participant inappropriate for the study.
* Positive pregnancy test for females of childbearing potential.
* Breastfeeding and childbearing potential female unwilling/unable to use a highly effective contraception method for the study duration and for at least 35 days after the last dose of lorlatinib
* Fertile male patients unwilling/unable to use a highly effective method of contraception for the duration of the study and for at least 97 days after the last dose of lorlatinib.
* Patients participating in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
* Patients deprived of their liberty, under protective custody or guardianship or unable to provide signed consent.
* Patients not affiliated to the French social security system.
* Patients opposed to the collection of their data.
* Patients willing and able to comply with the protocol for the duration of the study including undergoing treatment, scheduled visits and examinations including follow-up.
* Patients judged inapt to respond to the questions required for the study due to linguistical, psychological, social, or geographical reasons.
* Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From time of Study Start up to 25 months
  Time from inclusion to date of disease progression or death of any cause whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | From time of Study Start up to 25 months
  Time from inclusion to date of death from any cause.
Objective Response Rate (ORR) | From time of Study Start up to 24 months
  proportion of patients with a Complete Response (CR) or Partial Response (PR) as a best response during the lorlatinib treatment. Responses to treatment will be defined according to investigator
Duration of Response (DR) | From time of Study Start up to 24 months
  time between the first documentation of objective response and the first documentation of disease progression or death from any cause whichever occurred first, for participants with a confirmed objective response of CR or PR.
Intracranial Objective Response Rate (IC-ORR) | From time of Study Start up to 24 months
  proportion of patients with intracranial objective response of complete response (CR) or partial response (PR) as a best response in the subset of patients with at least 1 intracranial lesion assessed by investigator.
Intracranial Time to Progression (IC-TTP) | From time of Study Start up to 24 months
  Time from inclusion to the date of the first documentation of disease progression of intracranial disease, based on either new brain metastases or progression of existing brain metastases.
Intracranial Duration of Response (IC-DR) | From time of Study Start up to 24 months
  time from the first documentation of intracranial OR to the first documentation of intracranial progressive disease (PD) or death due to any cause, whichever occurred first for participants with a confirmed objective response of CR or PR assessed by investigator.
Duration of Treatment (DT) | From time of Study Start up to 25 months
  Time between inclusion and last dose of lorlatinib.
Proportion of patients with extracranial progression and sites of progression | From time of Study Start up to 24 months
  Based on Investigator's Assessment
Time to Treatment Failure (TTF) | From time of Study Start up to 24 months
  Time from date of treatment initiation to date of discontinuation of treatment for any reason, including progression of disease, treatment toxicity, and death from any cause whichever occurs first.
Adverse Event (AE) as graded by NCI CTCAE v5) | From time of Study Start up to 25 months
  Frequency of patients experiencing treatment-emergent AEs (TEAEs)
Number of Participants With Treatment-Emergent Adverse Events (AEs; Treatment-Related | From time of Study Start up to 25 months
  Treatment-emergent AEs were those with initial onset or that worsen in severity after the first dose of study medication. Treatment-related AEs were determined by investigators.
Proportion of patients considered observant to treatment assessed by the compliance questionnaire. | At the start of cycle (each cyle is 28 days) Cycle2Day1, Cycle3Day1, Cycle4Day1 and then every 3 months - as long as 48 months
  Self-administered questionnaire that provides a measure of compliance
Proportion of patients experiencing a 10-points change from baseline in total score for the EORTC QLQ-C30 | At inclusion, At the start of Cycle (each cycle is 28 days) Cycle2Day1, Cycle3Day1, Cycle4Day1 and every 3 months until the first year and then every 6 months - as long as 48 months
  evaluate Health-related Quality of life (HRQoL) of ALK- positive locally advanced or metastatic NSCLC patients treated with lorlatinib in first-line using the EORTC QLQ-C30 questionnaires
Proportion of patients experiencing a 10-points change from baseline in total score for the EORT QLQ-LC13. | At inclusion, At the start of Cycle (each cycle is 28 days) Cycle2Day1, Cycle3Day1, Cycle4Day1 and every 3 months until the first year and then every 6 months - as long as 48 months
  Evaluate Health-related Quality of life (HRQoL) of ALK- positive locally advanced or metastatic NSCLC patients treated with lorlatinib in first-line using the EORTC QLQ -LC13 questionnaires
Patient Reported Outcome-informed CNS symptomatic toxicity: | At inclusion, At the start of cycle (each cycle is 28 days) Cycle1Day15, Cycle2Day1, Cycle3Day1, Cycle4Day1 and every 3 months until the first year and then every 6 months - as long as 48 months
  frequency, severity and/or interference with daily activities, amount, presence/absence according to PRO-CTCAE questionnaires for mood (anxious/discouraged/sad), and attention/memory items (concentration/memory).
Proportion of patients experiencing grade III toxicities or progression and having an over- or under-exposure to lorlatinib. | At baseline, at start of Cycle1Day15 (each cycle is 28 days), Month 3, Month 9 and every 6 months through the end of treatment, at time of first grade III of hyperlipidaemia and CNS toxicity onset, and at progression - as long as 48 months
  At each time point, a blood sample to provide plasma for determination of the plasma concentrations of lorlatinib.
Proportion of patients experiencing each kind of identified lorlatinib resistance mechanisms | At baseline and at the date of first documented progression (as long as 48 months)
  Plasma samples collected at baseline and end of treatment, analyzed by next-generation sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Institut Godinot, Reims, France

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7461051